CLINICAL TRIAL: NCT05341115
Title: An Open Label, Multicenter, Single-arm and Prospective Study to Assess the Efficacy and Safety of Leuprorelin 3M in the Treatment of Central Precocious Puberty (CPP)
Brief Title: A Study of Leuprolide Acetate Depot in Children With Central Precocious Puberty
Acronym: PUPIL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Leuprorelin-4002; 2022-002471-11 (EudraCT Number)
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Central Precocious Puberty
Keywords: Drug Therapy
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Leuprorelin Acetate Depot 3M 11.25 mg (Experimental): Participants with CPP having body weight greater than equal to (≥)20 kilograms (kg) received the recommended dose of leuprorelin acetate depot 11.25 milligrams (mg) subcutaneous administration (SC) every 12 weeks based on the standard of 30～180 micrograms (μg)/kg/4 weeks for the 24-week Treatment Period. It was not recommended to exceed the dose above 180 μg/kg.
  Interventions: Drug: Leuprorelin Acetate Depot 3M

INTERVENTIONS:
Drug: Leuprorelin Acetate Depot 3M — Leuprorelin Acetate Depot 3M SC injections.
  Other Names: Leuprolide acetate Depot 3M

SUMMARY:
The main aim is to see how leuprolide works to treat central precocious puberty in children. Participants will receive an injection of leuprorelin acetate depot 11.25 mg every 12 weeks during 6 months and will visit their study clinic 6 times to complete some assessments.

DETAILED DESCRIPTION:
The drug being tested in this study is called leuprorelin acetate depot 3M. Leuprorelin acetate depot 3M will be tested to treat children who have central precocious puberty. This study will look at the efficacy and safety of leuprorelin acetate depot 3M in the treatment of CPP.

The study will enroll approximately 80 participants with CPP. Participants with a bodyweight of ≥ 20 kg will receive the recommended dose of leuprorelin acetate depot 3M in a 24 weeks Treatment Period followed by a 12 weeks Post-treatment follow-up period. Participants will be assigned to the following drug administration:

• Leuprorelin Acetate Depot 3M 11.25 mg

Participants will receive leuprorelin acetate depot 3M 11.25 mg as subcutaneous (SC) injection on Weeks 0, 12, and 24. The gonadotropin-releasing hormone agonist (GnRHa) stimulation, basal luteinizing hormone (LH), and follicle-stimulating hormone (FSH) levels will be tested pre-dose of every SC injection of the study drug or at premature termination.

This multi-center trial will be conducted in China. The overall time to participate in this study is 38 weeks. Participants will make a follow-up visit to the site at approximately 12 weeks after the last dose of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Maximum age to participate is this study is up to 10 years (child). Early appearance of secondary sexual characteristics: Girls ≤8 years, Boys ≤9years
2. Body weight ≥20 kg
3. According to the National Consensus Statement in China (2015), CPP is diagnosed when secondary sexual characteristics appeared before the age of 8 years in girls and 9 years in boys, a peak LH level >5.0 IU/L with LH/FSH >0.6 in stimulating test; evidence of gonadal development by ultrasonography (multiple ovarian follicles ≥4 mm in any ovary or uterine enlargement in females or testicular volume ≥4 mL in males); advanced bone age (BA) ≥1 year; linear growth acceleration with higher growth velocity (GV) than normal children. BA is determined by Greulich and Pyle standards or TW3 standards at screening.

Exclusion Criteria:

1. The participant has received GnRHa treatment in a previous clinical study or as a therapeutic agent.
2. The participant has a history or clinical manifestations of significant adrenal or thyroid diseases or intracranial tumor OR has a history of malignant disease.
3. The participant has a history of hypersensitivity or allergies to leuprorelin, or related compounds including any excipients of the compound.
4. The participant has a diagnosis of peripheral precocious puberty.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2025-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- China (5):
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - the First A liated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Hospital attached by the Torigji Medical College, Huazhong Science and Technology University., Wuhan, Hubei
  - Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Shanghai Children's Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/137c315e3a744cda?idFilter=%5B%22Leuprorelin-4002%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 79 participants took part in the study at 5 investigative sites in China from 14 March 2023 to 10 March 2025.
Pre-assignment Details: Participants with a diagnosis of central precocious puberty (CPP) received leuprorelin acetate depot 11.25 milligrams (mg).
Groups:
- Leuprorelin Acetate Depot 3M 11.25 mg: Participants with CPP having body weight greater than equal to (≥)20 kilograms (kg) received the recommended dose of leuprorelin acetate depot 11.25 mg subcutaneous administration (SC) every 12 weeks based on the standard of 30～180 micrograms (μg)/kg/4 weeks for the 24-week Treatment Period. It was not recommended to exceed the dose above 180 μg/kg.
Period: Overall Study
Arm/Group | Leuprorelin Acetate Depot 3M 11.25 mg
Started | 79
Completed | 77
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: The enrolled population set included all the eligible participants enrolled in this study, i.e., all participants enrolled in this study who met the inclusion criteria and did not meet any of the exclusion criteria, regardless of whether they received the study drug.
Groups:
- Leuprorelin Acetate Depot 3M 11.25 mg: Participants with CPP having body weight ≥20 kg received the recommended dose of leuprorelin acetate depot 11.25 mg SC every 12 weeks based on the standard of 30～180 μg/kg/4 weeks for the 24-week Treatment Period. It was not recommended to exceed the dose above 180 μg/kg.
Arm/Group | Leuprorelin Acetate Depot 3M 11.25 mg
Number analyzed (Participants) | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.59 (1.019)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 79
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 79
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Peak Luteinizing Hormone (LH) Suppression in Gonadotropin-Releasing Hormone (GnRH) Stimulation at Week 24
Description: The LH suppression was defined as LH peak value in GnRH stimulation ≤3.0 international unit per liter (IU/L).
Time Frame: Week 24
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprorelin Acetate Depot 3M 11.25 mg
Number analyzed (Participants) | 79
percentage of participants | 97.47 [91.15 to 99.69]

2. Secondary Outcome: Percentage of Participants With Tanner Stage Regression or No Progression at Week 24
Description: Tanner Stage was used to measure pubertal development. Tanner Stage was based on progression through 5-stages. The progression was defined as either breast/genitals or pubic hair score had increased score compared with baseline score. Otherwise, the status was classified as regression or no progression. Baseline is defined as the assessment prior to the first dose of study drug.
Time Frame: Baseline and Week 24
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprorelin Acetate Depot 3M 11.25 mg
Number analyzed (Participants) | 79
percentage of participants
  Tanner Stage Regression or No Progression | 97.47 [91.15 to 99.69]
  Tanner Stage Regression | 32.91 [22.75 to 44.40]
  No Tanner Stage Progression | 64.56 [52.99 to 75.00]

3. Secondary Outcome: Concentrations of Basal Luteinizing Hormone (LH) and Follicle Stimulating Hormone (FSH)
Description: Plasma LH and FSH peak concentrations under GnRH stimulation were assessed.
Time Frame: Baseline, Weeks 24 and 36
Population: The enrolled population set included all the eligible participants enrolled in this study, i.e., all participants enrolled in this study who met the inclusion criteria and did not meet any of the exclusion criteria, regardless of whether they received the study drug. Number analyzed is the number of participants with data available for analysis at the specified timepoints.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Leuprorelin Acetate Depot 3M 11.25 mg
Number analyzed (Participants) | 79
IU/L
  LH: Baseline: number analyzed (Participants) | 67
  LH: Baseline | 1.224 (1.410)
  LH: Week 24: number analyzed (Participants) | 70
  LH: Week 24 | 0.454 (0.297)
  LH: Week 36: number analyzed (Participants) | 75
  LH: Week 36 | 0.458 (0.293)
  FSH: Baseline | 3.213 (1.593)
  FSH: Week 24: number analyzed (Participants) | 75
  FSH: Week 24 | 1.457 (0.686)
  FSH: Week 36: number analyzed (Participants) | 77
  FSH: Week 36 | 1.569 (0.706)

4. Secondary Outcome: Percentage of Participants With Decreased Ratio of Bone Age Over Chronological Age at Week 24
Description: Bone age was determined by Greulich and Pyle standards or Tanner-Whitehouse 3 (TW3) standards.
Time Frame: Baseline and Week 24
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprorelin Acetate Depot 3M 11.25 mg
Number analyzed (Participants) | 79
percentage of participants | 84.81 [74.97 to 91.90]

5. Secondary Outcome: Percentage of Participants With Decreased First Morning Voided (FMV) Urinary Gonadotropin (Gn) at Week 24
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprorelin Acetate Depot 3M 11.25 mg
Number analyzed (Participants) | 79
percentage of participants
  Decrease in FMV Gn Urinary LH Values: number analyzed (Participants) | 74
  Decrease in FMV Gn Urinary LH Values | 62.03 [50.41 to 72.72]
  Decrease in FMV Gn Urinary FSH Values: number analyzed (Participants) | 78
  Decrease in FMV Gn Urinary FSH Values | 63.29 [51.69 to 73.86]

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. TEAE is defined as an AE with an onset that occurs after receiving study drug.
Time Frame: From first dose of study drug up to 12 weeks post last dose or early termination Visit (ET) (up to approximately 36 weeks)
Population: The safety population set included all included participants who had been under treatment with leuprorelin or who were first prescribed leuprorelin, received at least one dose and completed one follow-up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Leuprorelin Acetate Depot 3M 11.25 mg
Number analyzed (Participants) | 79
Participants | 27

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 12 weeks post last dose or early termination Visit (ET) (up to approximately 36 weeks)
Description: The safety population set included all included participants who had been under treatment with leuprorelin or who were first prescribed leuprorelin, received at least one dose and completed one follow-up visit.
Arm/Group | Leuprorelin Acetate Depot 3M 11.25 mg
All-Cause Mortality (participants affected / at risk) | 0/79
Serious Adverse Events (participants affected / at risk) | 1/79
Other Adverse Events (participants affected / at risk) | 4/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leuprorelin Acetate Depot 3M 11.25 mg (N=79)
Acute Appendicitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leuprorelin Acetate Depot 3M 11.25 mg (N=79)
Upper respiratory tract infection (Infections and infestations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-05-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT05341115/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT05341115/SAP_001.pdf